CLINICAL TRIAL: NCT01779193
Title: A Double-blind,Randomized,Parallel,Placebo-controlled Study of Probiotics Capsule as Supplemental Therapy for Group B Streptococci Infection and Vaginitis During Pregnancy
Brief Title: Probiotics Capsule as Supplemental Therapy for Group B Streptococci Infection and Vaginitis During Pregnancy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meng-Hsing Wu (Other)
Collaborators: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor-Investigator, Meng-Hsing Wu, National Cheng Kung University Hospital (NCKUH) Department of Obstetrics and Gynecology, National Cheng-Kung University Hospital
Organization: National Cheng-Kung University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A-BR-101-065
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Pregnancy
Keywords: group B streptococcus; pregnancy; probiotics
MeSH Terms: interventions — Lacteol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- latic acid bacteria and cranberry (Experimental): oral latic acid bacteria and cranberry capsule (dose of 2 * 10^9 cfu per capsule), one pill daily
  Interventions: Dietary Supplement: lactic acid bacteria; Dietary Supplement: cranberry
- cranberry (Active Comparator): oral cranberry capsule without lactic acid bacteria, one pill daily
  Interventions: Dietary Supplement: cranberry
- placebo (Placebo Comparator): placebo without lactic acid bacteria and cranberry, one pill daily
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: lactic acid bacteria — oral lactobacillus capsule (dose of 2 * 10^9 cfu per capsule), one pill daily
  Arms: latic acid bacteria and cranberry
Dietary Supplement: cranberry — oral cranberry capsule, one pill daily
  Arms: cranberry; latic acid bacteria and cranberry
Dietary Supplement: placebo — placebo capsule without lactic acid bacteria and cranberry, one pill daily
  Arms: placebo

SUMMARY:
B streptococcal infection and the major cause of death before and after the baby is born. B streptococcus infection the way of the newborn, usually infection from the mother in childbirth, if the pregnant women during pregnancy early diagnosis B streptococcus infection, it can be effective in preventing the risk of neonatal infection. Department of Health in China has been since April 15, 2012, the Scholarship holder at all pregnant women in the 35-37 weeks of pregnancy comprehensive B streptococcus screening. Infection B Streptococcus pregnant women in the labor process, the use of prophylactic antibiotics can be effective in reducing neonatal B streptococcus infection, but the possibility of the fetus being infected for the condition of premature birth or early rupture of membranes are still unable to fully hedge. In this study, the 35 to 37 weeks gestation examination confirmed infected B Streptococcus pregnant women, oral lactobacillus capsules B streptococcus infection treatment efficacy and safety assessment of clinical research. To assess whether oral administration of lactic acid bacteria will affect vaginitis incidence.

DETAILED DESCRIPTION:
Deeply influenced of bacterial vaginosis infection during pregnancy for pregnant women and fetus during childbirth, in which Group B Streptococcus agalactiae(GBS) is generally about 30% of pregnant women will be infected, about 1% vertical and infect the fetus, babies are not infected about 50% of the mortality rate in the treatment status, is considered an important reason for infection and death before and after the baby is born. Vertically in the natural childbirth process and infect the fetus, the delay in treatment on the fetus often lead to serious complications, including sepsis, pneumonia and meningitis, a serious will to cause death and permanent neurological sequelae, if given to confirm the diagnosis antibiotic treatment of pregnant women, the probability of infection of the newborn B streptococcus can be reduced by 75%. U.S. Centers for Disease Control recommends that pregnant women 35 to 37 weeks gestation or less than 37 weeks preterm contractions or rupture of membranes. B streptococcus check preterm doubts should pregnant women in the labor process and the use of preventive antibiotics can be effective in reducing neonatal B streptococcus infection, but the condition of premature birth or early rupture of membranes can not fully prevent the possibility of the fetus being infected is still in pre-production will not make any disposal, can cause infection of B The streptococci pregnant women worry, and under great pressure. This study for 35 to 37 weeks gestation to check to confirm infection of B Streptococcus pregnant women, pregnant women infected with the clinical studies of treatment efficacy and safety assessment of B streptococcus before delivery to the oral administration of lactic acid bacteria. The trial is expected during the execution in June 2012 to July 2015, subjects the number is expected to included at least 120 pregnant women choose not to subjects according to the conventional injection of prophylactic antibiotics in the labor process, choose to take oral lactobacillus oral lactobacillus of pregnant women in accordance with the 1:1 double-blind randomized to three groups, one of the following: test group A: oral lactobacillus capsules (dose of 2 x 109 cfu / capsule), experimental group B: oral without functional lactobacillus capsules and the control group: oral administration does not contain the active ingredient (lactic acid bacteria and cranberry) capsules before oral administration of lactic acid bacteria and the delivery process, collecting samples of vaginal anal secretions, whether positive addition to the screening B streptococcus, and the other selective medium coated plate culture for vaginal odor, itching number of the pathogen and B Streptococcus quantitative analysis and assessment questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* pregnancy women at 35 weeks of gestation

Exclusion Criteria:

* previous other probiotics capsules use
* previous antibiotics use
* previous habitual vaginal douche
* previous medical disease, such as: HIV infection, cancer, history of organ transplantation, long-term steroid use, autoimmune disease, et al

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-06; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
all cases vaginal group B streptococcus colonies | four years

CONTACTS AND LOCATIONS:
Overall Officials: Meng-Hsing Wu, M.D., Ph.D., Principal Investigator — National Cheng Kung University
Locations (1):
- Department of Obstetrics and Gynecology, College of Medicine, National Cheng Kung University, Tainan, Taiwan